CLINICAL TRIAL: NCT00904280
Title: An Open-Label Extension Study to Evaluate the Long-Term Safety, Tolerability and Analgesic Efficacy of Numorphan® CR (Oxymorphone HCL Controlled Release) in Subjects With Cancer Pain or Chronic Lower Back Pain.
Brief Title: Open-Label Extension to Evaluate the Long-Term Safety, Tolerability and Analgesic Efficacy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director, Cliniacal R&D, Endo Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3202-021
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2009-05-19 (Estimated); Status verified 2009-03

CONDITIONS: Cancers, Pain; Lower Back Pain
MeSH Terms: conditions — Neoplasms; Pain; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxymorphone ER (Experimental)
  Interventions: Drug: Oxymorphone ER

INTERVENTIONS:
Drug: Oxymorphone ER — Open label

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of oxymorphone ER as an analgesic in cancer and lower back pain subjects having chronic moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* The subject enrolled in this study must have been previously randomized and dosed in the double-blind treatment period of study EN3202-016 or EN3202-019 and completed the exit visits for these studies.
* Males or females, age 18 and 75 years, inclusively.
* The subject continues to have chronic moderate to severe back or cancer pain that requires opioid medication. Women must continue to be of non-childbearing potential.

Exclusion Criteria:

* The subject experienced any serious drug related adverse events in studies EN3202-016 or EN3202-019.
* The subject withdrew from EN3202-016 or EN3202-019 for a reason other than lack of efficacy.
* Subjects with known allergies to opiate-class narcotic agents (morphine, codeine, hydrocodone, propoxyphene, meperidine, oxycodone, etc.) or naproxen, or subjects who have any medical condition in which opiates are medically contraindicated.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2001-03; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Monthly assessments of pain with the Brief Pain Inventory (BPI) questionnaire, recall of average pain relief, total rescue medication usage and subject's and physician's global assessment of oxymorphone ER | 1 year study

SECONDARY OUTCOMES:
To evaluate long-term efficacy of oxymorphone ER as an analgesic in cancer and lower back pain subjects having chronic moderate to severe pain | 1 year study

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director, Study Director — Endo Pharmaceuticals
Locations (1):
- Arizona Clinical Research Center, Tucson, Arizona, United States